CLINICAL TRIAL: NCT05481099
Title: Efficacy of a Cognitive Behavioural-based Intervention in Reducing Test Anxiety in High School Students: a Pilot Cluster Randomized Controlled Trial
Brief Title: Reducing Test Anxiety in High School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agrupamento de Centros de Saúde de Dão Lafões (Other)
Collaborators: Casa de Saúde São Mateus - Hospital (Unknown)
Responsible Party: Principal Investigator, Frederico Rosário, MD, PhD, Head of Research Department, Agrupamento de Centros de Saúde de Dão Lafões
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Anxiety-2020
Record Dates: First submitted 2022-07-27; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Test Anxiety
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Cognitive-behavioural-based intervention combined with mindfulness, psychoeducation, and relaxation techniques
  Interventions: Behavioral: Intervention
- Control (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: Intervention — Cognitive-behavioural-based intervention combined with mindfulness (attention focus), psychoeducation, and relaxation techniques (short version of Jacobson's progressive relaxation, breathing exercises)
  Arms: Intervention

SUMMARY:
School-age test anxiety is an important risk factor for school performance. Notwithstanding, few studies seek to identify which strategies are effective in improving test anxiety. This study aimed to test whether a cognitive-behavioural intervention for high school students could significantly reduce test anxiety.

A two-arm, cluster-randomized controlled, unblinded, parallel, trial was conducted. Participants were students of the 10th year of the Alves Martins High School in Viseu, Portugal. Students were randomized at class level to receive a cognitive-behavioural-based intervention combined with mindfulness, psychoeducation, and relaxation techniques, or to a control group with no intervention. Participants' anxiety levels were measured using the Test Anxiety Questionnaire. The analysis of the effect of the intervention was carried out on an intention-to-treat basis at the class level, using multilevel mixed effects models and Bayesian modelling.

ELIGIBILITY:
Inclusion Criteria:

* 10th grade students; both students and parents provide written informed consent

Exclusion Criteria:

* cognitive inability to answer the questionnaire and/or to participate in the intervention

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Test anxiety | 12 weeks
  Participants' test anxiety will be assessed using the Test Anxiety Questionnaire. Scores on the questionnaire range from 10 to 50 points. Higher scores mean higher anxiety levels.

SECONDARY OUTCOMES:
Worry | 12 weeks
  Participants' worry will be assessed using the Worry subscale (items 1-5) of the Test Anxiety Questionnaire. Scores on the questionnaire range from 5 to 25 points. Higher scores mean higher worry-related anxiety levels.
Emotionality | 12 weeks
  Participants' emotionality will be assessed using the Emotionality subscale (items 6-10) of the Test Anxiety Questionnaire. Scores on the questionnaire range from 5 to 25 points. Higher scores mean higher emotionality-related anxiety levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Alves Martins High School, Viseu, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopes D, Ferrao A, Matanca AF, Almeida C, Rosario F, Santos J, Santos MI. [A Cognitive Behavioural-Based Intervention in Reducing Test Anxiety in High School Students: A Pilot Cluster Randomized Controlled Trial]. Acta Med Port. 2024 Feb 5;37(3):163-171. doi: 10.20344/amp.18876. Epub 2023 Mar 20. Portuguese. PMID 36939679